CLINICAL TRIAL: NCT05825742
Title: Efficacy of Regular Home Use of Dual-light Photodynamic Therapy on Oral Health in Adolescents Undergoing Fixed Orthodontic Treatment - Randomized, Controlled Clinical Study
Brief Title: Regular Home Use of Dual-light Photodynamic Therapy on Oral Health in Adolescents Undergoing Fixed Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Helsinki (Other); Helsinki University Central Hospital (Other); Borgska Villans Specialisttandvård (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEAN-BRACKET
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Orthodontic Appliance Complication; Plaque, Dental; Gingival Inflammation
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: Participants in two groups (Study group and Control group) shall receive instructions for standard oral hygiene. The same assessments are done for participants in both groups, and within the same time periods. The Study group will also be using the Lumoral Treatment device.
Masking Description: The participants, care providers, and investigators shall be masked before the first measurements. The randomization will be conducted after the first measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumoral Treatment (Study group) (Experimental): Subjects will receive detailed instructions for the use of Lumoral treatment -device. Subjects will be instructed to use the Lumoral treatment -device and follow the protocol once a day for two months and to keep a diary.
  Subjects will receive the latest standard oral hygiene instructions according to the Swedish dental association's guidelines.
  Interventions: Device: Lumoral Treatment; Other: Standard oral health instructions
- Standard of care (Control group) (Other): Subjects will receive the latest standard oral hygiene instructions according to the Swedish dental association's guidelines.
  Interventions: Other: Standard oral health instructions

INTERVENTIONS:
Device: Lumoral Treatment — Subjects will receive detailed instructions for the use of Lumoral treatment -device. Subjects will be instructed to use the Lumoral treatment -device and follow the protocol once a day for two months and to keep a diary.
  Arms: Lumoral Treatment (Study group)
Other: Standard oral health instructions — Subjects will receive the latest standard oral hygiene instructions according to the Swedish dental association's guidelines.

SUMMARY:
This study is designed to determine the efficacy of the Lumoral method on oral health in adolescents undergoing fixed orthodontic treatment. Improved supragingival plaque control can help to also sustain the subgingival plaque management in the long term. In addition, the device might have a photobiomodulation effect on periodontal tissues.

DETAILED DESCRIPTION:
Orthodontic treatment is one of the most common dental treatments in children and adolescents. The use of fixed orthodontic appliances makes it difficult for the patients to keep their oral hygiene to an optimum level of cleanliness. Poor oral hygiene attracts significant plaque accumulation around the fixed orthodontic treatment appliances, and subsequent white spot lesions can occur rapidly, usually on the cervical and middle third of the buccal surfaces of bracketed teeth. Patients with the fixed orthodontic treatment appliances have an increased risk of caries and gingivitis.

The Lumoral is a CE-marked medical device developed to provide a potent, targeted antibacterial action on dental plaque in a home environment. The device mechanism of action is antibacterial photodynamic therapy (aPDT). The device is used by swishing a mouth rinse, which has a strong adherence to dental plaque. The plaque-adhered photoactive mouth rinse can be activated by a simple to use light applicator. Preliminary results have shown a promising anti-inflammatory response in addition to plaque reduction.

Forty (40) subjects undergoing fixed orthodontic treatment are randomized to the Lumoral treatment group or the control group. All subjects shall receive polishing and oral hygiene instruction. All patients shall be assessed for the clinical measurements including visible plaque index (VPI), bleeding on probing (BOP), and orthodontic plaque index (OPI) at baseline and at 4 weeks and 12 weeks after baseline. In addition, microbiological analyses shall be performed at baseline and at 12 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* age of 15-18 years old
* starting fixed orthodontic treatment
* good oral hygiene according to the dentist's assessment
* absence of periodontal disease and lack of oral lesion
* signed a written consent form, including information to caregivers.

Exclusion Criteria:

* any chronic diseases
* medications that could influence the study (according to the dentists' assessment)
* active caries or a supposed high risk of caries
* gingivitis (bleeding on probing >10%)
* use of antiseptic mouthwashes
* smoking
* use of antibiotics or anti-inflammatory therapy within 3 months before entering the study or during the study
* unable to cooperate with the protocol.
* pregnancy or lactation

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Visible plaque index (VPI) | 12 weeks
  * A full-mouth assessment, measured at six sites per tooth.
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * VPI is reported as the percentage (%) of sites with plaque.
  * Calculation formula: number of sites with plaque/ 6 times number of teeth

SECONDARY OUTCOMES:
Change in Bleeding on probing (BOP) | 12 weeks
  * A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual)
  * Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus.
  * Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent"
  * BOP is reported as the percentage (%) of sites with positive findings.
  * Calculation formula: number of bleeding sites/ 6 times number of teeth
Change in Orthodontic plaque index (OPI) | 12 weeks
  * The OPI indicates the presence of plaque around the multibracket appliance after staining the teeth with a plaque-disclosing solution.
  * Using the data from the digital photographs, selected six (6) index teeth that bear an adhesively bonded bracket will be evaluated.
  * The status is indicated as a score from 0 to 4. The degree of plaque accumulation on each aspect of the bracket base and the condition of the adjacent marginal gingivae are assessed: 0 = No plaque deposits on the tooth surfaces surrounding the bracket base
    1. = Plaque deposits on one tooth surface at the bracket base
    2. = Plaque deposits on two tooth surfaces at the bracket base
    3. = Plaque deposits on three tooth surfaces at the bracket base
    4. = Plaque deposits on four tooth surfaces at the bracket base and/or gingival inflammation indicators (plaque deposits near the gingiva do not necessarily have to be present)
Change in periodontal microbiological flora | 12 weeks
  Microbiological sampling and analysis:
  * Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis.
  * Microbiological samples can be collected using Iso Taper Paper Points, size-20 (VDW GmbH) from the plaque on the surface of the teeth, using a curette if needed. The paper points can be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis.
  * 16S rRNA sequencing can be performed at a qualified laboratory assigned by the study sponsor

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Roos Jansåker, Professor, Principal Investigator — Borgska Villans Specialisttandvård; Tommi Pätilä, Docent, Study Director — Koite Health
Locations (1):
- Borgska Villans Specialisttandvård, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erbe C, Klees V, Braunbeck F, Ferrari-Peron P, Ccahuana-Vasquez RA, Timm H, Grender J, Cunningham P, Adam R, Wehrbein H. Comparative assessment of plaque removal and motivation between a manual toothbrush and an interactive power toothbrush in adolescents with fixed orthodontic appliances: A single-center, examiner-blind randomized controlled trial. Am J Orthod Dentofacial Orthop. 2019 Apr;155(4):462-472. doi: 10.1016/j.ajodo.2018.12.013. PMID 30935601
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Verrusio C, Iorio-Siciliano V, Blasi A, Leuci S, Adamo D, Nicolo M. The effect of orthodontic treatment on periodontal tissue inflammation: A systematic review. Quintessence Int. 2018;49(1):69-77. doi: 10.3290/j.qi.a39225. PMID 29114647
- [Background] Walsh LJ, Healey DL. Prevention and caries risk management in teenage and orthodontic patients. Aust Dent J. 2019 Jun;64 Suppl 1:S37-S45. doi: 10.1111/adj.12671. PMID 31144319
- See also: Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review. Laser Dent Sci 3, 147-153 (2019) — https://link.springer.com/article/10.1007/s41547-019-00056-9
- See also: Levine JI. Medications that increase photosensititivity. FDA document Dec 1990. — https://www.fda.gov/media/75892/download
- See also: Linden J, Widström E & Sinkkonen J (2019) Children and adolescents´ dental treatment in 2001-2013 in the Finnish public dental service. BMC Oral Health (2019) 19:131 — https://bmcoralhealth.biomedcentral.com/articles/10.1186/s12903-019-0828-z
- See also: Nikinmaa S, Alapulli H, Auvinen P, et al. (2020) Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. PLoS ONE 15(5) — https://doi.org/10.1371/journal.pone.0232775
- See also: Pereira PAB, Aho VTE, Paulin L, et al., (2017) Oral and nasal microbiota in Parkinson's disease. Parkinsonism and Related Disorders 38: 61-67 — https://doi.org/10.1016/j.parkreldis.2017.02.026